CLINICAL TRIAL: NCT04559893
Title: Improving Access and Treatment for Co-occurring Opioid Use Disorders and Mental Illness
Brief Title: Collaboration Leading to Addiction Treatment and Recovery From Other Stresses
Acronym: CLARO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: University of New Mexico (Other); Boston Medical Center (Other); First Choice Community Healthcare (Unknown); Hidalgo Medical Services (Unknown); National Institute of Mental Health (NIMH) (NIH); Stanford University (Other); University of Pittsburgh (Other); Saint John's Cancer Institute (Other); Olive View-UCLA Education & Research Institute (Other)
Responsible Party: Principal Investigator, Katherine Watkins, Senior Physician Policy Researcher, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1UF1MH121954 (NIH); 1UF1MH121954 (NIH)
Record Dates: First submitted 2020-09-08; First posted 2020-09-23 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Opioid-use Disorder; Addiction; Depression; Post-traumatic Stress Disorder
Keywords: Collaborative care; Problem solving therapy; Written exposure therapy; Medication for addiction treatment; Addiction; Opioid-use disorder
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Two-arm randomized control trial (RCT) where participants are randomly assigned to intervention or control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative Care (Experimental): Intervention is administered to patients in this arm. Care to be delivered via collaborative care.
  Interventions: Behavioral: Collaborative Care
- Control (No Intervention): Patients in this arm will receive enhanced usual care.

INTERVENTIONS:
Behavioral: Collaborative Care — Collaborative care consists of a team of providers that includes a care coordinator, a primary care provider (PCP) and a behavioral health consultant (BHC), who provide evidence- and measurement-based care to a panel of patients using a clinical registry. In our model, the CC team also includes a behavioral health psychotherapist (BHP) who consults on a regular basis but does not deliver direct care.
  Arms: Collaborative Care

SUMMARY:
Collaboration Leading to Addiction Treatment and Recovery from Other Stresses (CLARO) is a five-year project that tests whether delivering care using a collaborative model helps patients with both opioid use disorders and mental health disorders.

DETAILED DESCRIPTION:
Untreated mental illness and substance use disorders are prevalent and can have devastating consequences for the individual, their families and the community. Co-occurring opioid use disorders (OUD) with either depressive disorders and/or post-traumatic stress disorder (PTSD) are of particular concern, because depression and PTSD are prevalent in people with OUD, co-occurring mental illness is linked to an increased risk for opioid misuse and overdose, and because of the high prevalence of the chronic use of prescription opioids in individuals with mental illness, a risk factor for heroin use and the development of an OUD. Primary care is an important and underutilized setting in which to provide treatment for all three disorders, because OUD, depression and PTSD are frequently co-morbid with medical conditions. However, despite the effectiveness of treatments for all three disorders, many individuals never receive treatment; and, when treatment is provided, quality is low. With the rising number of opioid-related fatalities, this is a critical treatment and quality gap in a vulnerable and stigmatized population. Collaborative care (CC) has never been tested with co-occurring disorders (COD), despite research by our team suggesting it may be effective. CC consists of a team of providers that includes a care coordinator, a primary care provider (PCP) and a behavioral health consultant (BHC), who provide evidence- and measurement-based care to a panel of patients using a clinical registry. In our CC model for COD (CC-COD), the CC team also includes a behavioral health psychotherapist (BHP); the evidence-based treatments supported include medications for OUD (MOUD), pharmacotherapy for depression and PTSD, motivational interviewing (MI), problem solving therapy (PST) and Written Exposure Therapy (WET).

The current study consists of a multi-site, randomized pragmatic trial in rural and urban primary care clinics located in Health Professional Shortage Areas (HPSA) of New Mexico and California to adapt, harmonize and then test whether CC-COD improves access, quality and outcomes for primary care patients with co-morbid OUD and depression and/or PTSD. The study will randomize 900 patients with co-occurring OUD and depression disorder and/or PTSD to receive either CC-COD or enhanced usual care (EUC).

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Receiving primary care at one of the participating clinical sites
* Has OUD and one or more specific co-occurring behavioral health disorders (depression and PTSD)

Exclusion Criteria:

* Under 18
* Does not speak English or Spanish
* Unable to consent
* Receiving both MOUD and psychotropic medication from a provider outside of the primary care health system at which the patient is enrolled
* Not receiving primary care at one of the participating clinical sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 729 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Buprenorphine access | Assessed at 6 months after study entry.
  Number of days until first buprenorphine prescription after study enrollment for study participants with a new episode of OUD care (no care for at least 30 days prior). Obtained from the Prescription Drug Monitoring Program and patient survey.
Buprenorphine continuity of care | Assessed at 6 months after study entry.
  The cumulative number of days the patient receives buprenorphine during the 180 days after study enrollment for study participants not on methadone at baseline. Obtained from the Prescription Drug Monitoring Program and patient survey.
Major Depressive Disorder (MDD) symptom severity | Assessed at 6 months after study entry.
  Sum of items (0-27) in the PHQ-9 (Patient Health Questionnaire) at 6 months for participants with probable major depression at baseline.
Post-traumatic Stress Disorder (PTSD) symptom severity | Assessed at 6 months after study entry.
  Sum of items (0-80) in PCL-5 at 6 months for study participants with probable PTSD at baseline.

SECONDARY OUTCOMES:
Access to MDD and/or PTSD treatment | Assessed at 30 days and 180 days after study entry.
  Receipt of medication and/or behavioral treatment associated with an MDD or PTSD diagnosis within 30 days of study enrollment (initial) or within 180 days of study enrollment (any) for study participants who did not have any visits (behavioral health treatment or medication) for MDD and/or PTSD in 30 days prior to study enrollment. Obtained from patient survey and electronic medical records.
Quality of care for MDD | Assessed at 6 months after study entry.
  Four psychotherapy visits in the first six months or an adequate (60 day) medication trial for new episodes of MDD care (completed within 6 months) for study participants with probable MDD at baseline and a new episode of MDD care (no MDD care for at least 30 days prior to enrollment). Obtained from patient survey and electronic medical records.
Quality of care for PTSD | Assessed at 6 months after study entry.
  Four psychotherapy visits in the first six months or an adequate (60 days) medication trial for new episodes of PTSD care (completed within 6 months) for study participants with probable PTSD at baseline, and a new episode of PTSD care (no PTSD care for at least 30 days prior to enrollment). Obtained from patient survey and electronic medical records.
MDD remission | Assessed at 6 months after study entry
  Binary measure based on sum of items (0-27) in the PHQ-9. PHQ-9 score less than 5 at 6 months for study participants with probable MDD at baseline.
MDD response | Assessed at 6 months after study entry.
  Binary measure based on sum of items (0-27) in the PHQ-9. PHQ-9 score at 6 months less than 50% of baseline score for participants with probable MDD at baseline.
PTSD remission | Assessed at 6 months after study entry.
  Binary measure based on sum of items (0-80) in the PCL-5. PCL-5 score less than 34 at 6 months for study participants with probable PTSD at baseline.
PTSD response | Assessed at 6 months after study entry.
  Binary measure based on sum of items (0-80) in the PCL-5. PCL-5 score at 6 months less than 50% of baseline score for study participants with probable PTSD at baseline.
Active suicidal ideation | Assessed at 6 months after study entry.
  Dichotomized Columbia Suicide Severity Rating Scale at 6 months. Endorsed if participants answer YES to Question 3, 4, and/or 5 and/or YES to Question 7. Obtained from patient survey.
Opioid use frequency | Assessed over 30 days after study entry.
  Days of opioid use in the past 30 days from National Survey on Drug Use and Health. Obtained from patient survey.
Opioid overdose events | Assessed over the previous 3 months after study entry.
  Opioid overdose events (at least 1 event) in the previous three months. Obtained from patient survey.
Physical health functioning | Assessed at 30 days after study entry
  Physical health measured using the component scores from the Veterans RAND 12-item Health Survey (VR-12) physical health subscale.
Mental health functioning | Assessed at 30 days after study entry
  Mental health functioning measured using the component scores from the Veterans RAND 12-item Health Survey (VR-12) mental health subscale.

OTHER OUTCOMES:
Drug use frequency | Assessed over 30 days after study entry.
  Maximum days of use in the past 30 days for five drug categories using items from National Survey on Drug Use and Health (prescription opioids, heroin, cocaine/crack, methamphetamine/ other stimulants, and tranquilizers/sedatives). Obtained from patient survey.
Stimulant use frequency | Assessed over 30 days after study entry.
  Days of stimulant use (cocaine/crack, methamphetamine/ other stimulants) in the past 30 days from the National Survey on Drug Use and Health. Obtained from patient survey.
Alcohol use | Assessed over 3 months after study entry.
  Sum of items (0-12) in the Alcohol Use Disorder Identification Test - Consumption (AUDIT-C) for the previous 3 months.
Opioid overdose risk behaviors | Assessed over 3 months after study entry.
  Sum of 32-items in the Opioid Overdose Risk Assessment.
Opioid use severity | Assessed over 30 days after study entry.
  Sum of items (7-35) in the Patient-Reported Outcomes Measurement Information System (PROMIS) Substance Use Short Form for the previous 30 days. Obtained from patient survey.
Demographics | Assessed at study entry.
  Self-reported demographics on age, sex, race/ethnicity, educational attainment, and marital status.
Pain levels | Assessed over the previous 7 days at study entry and at 3 and 6 months after study entry
  Pain Intensity, Enjoyment of Life, General Activity (PEG) Pain Monitor for the past week; assessed as a covariate; obtained from patient interview
History of MOUD treatment | Asked about lifetime MOUD treatment; assessed at study entry
  Assessed as a covariate; obtained from patient interview
Current MDD/PTSD treatment | Assessed over the previous 30 days at study entry
  NSDUH items; assessed as a covariate; obtained from patient interview
Prior experience with a care coordinator | Assessed over the previous 12 months at study entry
  Assessed as a covariate; obtained from patient interview
Homelessness | Assessed over the previous 3 months at study entry
  Homelessness Screening Clinical Reminder Tool and one item from the Government Performance and Results Act (GPRA) clarifying where individuals who are homeless are currently living; assessed as a mediator; obtained from patient interview
Disability and impairment | Assessed over the previous 7 days at study entry
  3-item Sheehan Disability Scale; assessed as a covariate; obtained from patient interview
Clinician (care coordinator) communication | Assessed over the previous 3 months at 3 months after study entry
  Agency for Healthcare Research and Quality (AHRQ) Consumer Assessment of Healthcare Providers and Systems survey items; assessed as a mediator; obtained from patient interview
Ability to access treatment quickly | Assessed over the previous 3 months at 3 months after study entry
  AHRQ Consumer Assessment of Healthcare Providers and Systems survey items; assessed as a mediator; obtained from patient interview
Satisfaction with treatment | Assessed over the previous 3 months at 3 months after study entry
  AHRQ Consumer Assessment of Healthcare Providers and Systems survey items; assessed as a mediator; obtained from patient interview
Patient-care manager working alliance | Assessed over the previous 3 months at 3 months after study entry
  Modified Working Alliance Inventory-General Practitioner (WAI-GP); assessed as a mediator; obtained from patient interview

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Watkins, Principal Investigator — RAND; Miriam Komaromy, Principal Investigator — Boston Medical Center
Locations (16):
- United States (16):
  - Hubert Humphrey Comprehensive Health Center, Los Angeles, California
  - Providence Saint John's Health Center, Santa Monica, California
  - First Choice Community Healthcare - South Broadway Medical Center, Albuquerque, New Mexico
  - First Choice Community Healthcare - South Valley Medical/Dental Center, Albuquerque, New Mexico
  - First Choice - Alameda Medical Center, Albuquerque, New Mexico
  - First Choice Community Healthcare - North Valley Medical Center, Albuquerque, New Mexico
  - University of New Mexico Family Health Clinic, North Valley, Albuquerque, New Mexico
  - University of New Mexico Family Health Clinic, Southeast Heights, Albuquerque, New Mexico
  - First Choice Community Healthcare - Alamosa Medical Center, Albuquerque, New Mexico
  - University of New Mexico Internal Medicine Clinic, Southwest Mesa, Albuquerque, New Mexico
  - First Choice Community Healthcare - Belen Medical Center, Belen, New Mexico
  - First Choice Community Healthcare - Edgewood Medical/Dental Center, Edgewood, New Mexico
  - Hidalgo Medical Services - Lordsburg Clinic, Lordsburg, New Mexico
  - First Choice Community Healthcare - Los Lunas Medical/Dental Center, Los Lunas, New Mexico
  - Hidalgo Medical Services - Community Health Center, Silver City, New Mexico
  - Hidalgo Medical Services - Med Square Clinic, Silver City, New Mexico

IPD SHARING:
Plan to Share IPD: Yes
Per National Institute of Mental Health (NIMH) funding requirements, study data must be uploaded to the NIMH National Data Archive (NDA) every six months once data collection begins. A universal subject identifier called a Global Unique Identifier (GUID) will be generated for each participant. All raw data will be uploaded every six months to the NIMH NDA per their policies. Additionally, all analysis data sets used for manuscripts must be uploaded to the NIMH NDA, identified by GUID.
Time Frame: Every 6 months (January and July) following enrollment of the first patient. First submission expected July 2021. Submission will cease following sharing of final analysis data set for any specified outcomes publications.
Access Criteria: Per NIMH NDA policies (https://nda.nih.gov/)
URL: https://nda.nih.gov/

REFERENCES:
- [Derived] Watkins KE, Osilla KC, McCullough CM, Griffin BA, Dopp AR, Becker K, Meredith LS, Carrejo V, Hindmarch GM, Mendon-Plasek S, Christensen J, Weir R, Kelly L, Pak L, Murray-Krezan C, Tarhuni L, Crowley C, Bilder A, Kalmin MM, Schoenbaum M, Komaromy M. Collaborative Care for Opioid Use Disorder and Mental Illness: The CLARO Randomized Clinical Trial. JAMA Intern Med. 2025 Dec 29:e257036. doi: 10.1001/jamainternmed.2025.7036. Online ahead of print. PMID 41460640
- [Derived] Hindmarch G, Meredith LS, McCullough CM, Griffin BA, Watkins KE. Interpersonal Violence and Mental Health, Drug use, and Treatment Utilization among Patients with Co-Occurring Opioid use and Mental Health Disorders. Chronic Stress (Thousand Oaks). 2024 Sep 5;8:24705470241279335. doi: 10.1177/24705470241279335. eCollection 2024 Jan-Dec. PMID 39246736
- [Derived] Osilla KC, Meredith LS, Griffin BA, Martineau M, Hindmarch G, Watkins KE. Design of CLARO+ (Collaboration Leading to Addiction Treatment and Recovery from Other Stresses, Plus): A randomized trial of collaborative care to decrease overdose and suicide risk among patients with co-occurring disorders. Contemp Clin Trials. 2023 Sep;132:107294. doi: 10.1016/j.cct.2023.107294. Epub 2023 Jul 16. PMID 37454728
- [Derived] Osilla KC, Dopp AR, Watkins KE, Ceballos V, Hurley B, Meredith LS, Leamon I, Jacobsohn V, Komaromy M. Collaboration Leading to Addiction Treatment and Recovery from Other Stresses (CLARO): process of adapting collaborative care for co-occurring opioid use and mental disorders. Addict Sci Clin Pract. 2022 Apr 8;17(1):25. doi: 10.1186/s13722-022-00302-9. PMID 35395811

DOCUMENTS (3):
  • Study Protocol (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT04559893/Prot_002.pdf
  • Statistical Analysis Plan (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT04559893/SAP_003.pdf
  • Informed Consent Form (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT04559893/ICF_000.pdf